CLINICAL TRIAL: NCT06163183
Title: The Potential of Diaphragm Electrical Activity Monitoring to Predict Extubation Success in Children Requiring Mechanical Ventilation Support Due to Respiratory Failure
Brief Title: Does Diaphragm Electrical Activity Monitoring Predict Extubation Success in Children?
Status: Completed | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Edanur Yesil, MD, Associate Professor, Mersin University
Other Study IDs: 1400124188
Record Dates: First submitted 2023-11-27; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Diaphragm Electrical Activity; Neurally Adjusted Ventilatory Assist; Pediatrics
Keywords: pediatrics; extubation success; Diaphragm electrical activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Extubation failure
  Interventions: Device: Edi catheter
- Extubation success
  Interventions: Device: Edi catheter

INTERVENTIONS:
Device: Edi catheter

SUMMARY:
This study aimed to record diaphragm electrical activity (Edi) during the preextubation (weaning) and postextubation periods and to analyze whether Edi monitoring could predict extubation success.

DETAILED DESCRIPTION:
This prospective observational study included 25 pediatric patients who were intubated due to respiratory failure in the pediatric intensive care unit of the tertiary university-affiliated Marmara University Hospital between August 2014 and July 2015. To conduct the study, we obtained informed consent from the patient's parents and ethical approval from the Marmara University Faculty of Medicine Scientific Research Ethics Committee Board on 06.09.2014. Pediatric patients included which had indication for the insertion of a nasogastric tube (Edi catheter), independent of the study. So Edi catheter had been used instead of nasogastric tube.

When the patients were ready for clinical weaning in accordance with the clinician, the Edi catheter was appropriately inserted into the patients. Then, a spontaneous breathing trial (SBT) was performed and diaphragm activity monitoring was recorded during this process. The patients who met the inclusion criteria switched in a spontaneous breath trial with pressure support ventilation (PSV) or NAVA (Neurally Adjusted Ventilatory Assist) on a Maquet (Solna, Sweden) Servo-i mechanical ventilator for both ventilation modes The patients' demographic and clinical characteristics, mortality scoring, vital parameters (HR, TA, SpO2, RR) and ventilatory parameters (Edi peak, Edi min, FiO2, expiratory Vt), as well as follow-up period were recorded. Arterial/capillary blood gases were taken within the last four hours before extubation and within the first, sixth, 12th, 18th and 24th hours after extubation. If arterial blood gas monitoring was initiated in the patient, arterial monitoring was continued. If capillary blood gas monitoring was initiated, capillary monitoring was continued. Edi data were recorded for at least 24 hours before and after extubation. Edi values were obtained retrospectively from the trend diagram, which provides 24-hour continuous records on the ventilator screen.

ELIGIBILITY:
Inclusion Criteria:

* • Aged between one month and 18 years old

  * Intubated for more than 48 hours due to respiratory failure
  * Indication for the insertion of a nasogastric tube (Edi catheter), independent of the study
  * Ready for weaning:

    * Normal vital signs for age (fever, heart rate (HR), respiratory rate (RR), tension arterial (TA)
    * No catecholamines or sedation drugs
    * pH of 7.35 to 7.45
    * Positive end expiratory pressure (PEEP) ≤6 mmHg
    * Fractionated oxygen (FiO2) ≤0.5
    * Oxygen saturation (SpO2) ≥92%
    * Vt≥ 5 ml/kg

Exclusion Criteria:

* • Contraindication for the insertion of the nasogastric tube (Edi catheter)

  * Patients treated with muscle relaxants
  * Absence of consent given by the patient's family
  * Cases whose Edi levels could not be taken from ventilator's trend diagram due to missing values.

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The majority of the patients were under 18 months of age (median 18 months, between 2 and 204 months) and 60% (n=15) were female.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2015-07-30 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Diaphragm electrical activity (Edi) monitoring | up to 2 days
  Macquet (servo-i) mechanical ventilator measures the electrical activity (Edi) of the diaphragm (microvolts). Edi signals are measured using special feeding tubes (Edi catheter) equipped with tiny sensors at the level of gastroesophageal junction. In the ventilator, Edi trend values can be monitored continuously as 24-hour records.
Mechanical ventilatory monitoring | up to 2 days
  ventilatory parameters (Edi peak, Edi min, FiO2), were recorded during the follow up.

SECONDARY OUTCOMES:
Arterial/capillary blood gases | Arterial/capillary blood gases were taken within the last four hours before extubation and within the first, sixth, 12th, 18th and 24th hours after extubation.
  If arterial blood gas monitoring was initiated in the patient, arterial monitoring was continued. If capillary blood gas monitoring was initiated, capillary monitoring was continued.
Vital signs ((fever, heart rate (HR), respiratory rate (RR), tension arterial)) | up to 2 days
  Vital signs recorded by pediatric intensive care nurses.
Expiratory tidal volume | From spontaneous breathing trial until the time for extubation
  Patients who had >5ml/kg expiratory tidal volume considered to be ready for extubation

CONTACTS AND LOCATIONS:
Overall Officials: Nilufer Yalindag-Ozturk, Proffessor, Study Director — Marmara University Medical Faculty, Pediatric Intensive Care Speacilist

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, will be shared in publication study
Supporting Information: Study Protocol, SAP
Time Frame: 4 month
Access Criteria: After publication of study, the study will be shown by request.

REFERENCES:
- [Result] Beck J, Sinderby C. Neurally Adjusted Ventilatory Assist in Newborns. Clin Perinatol. 2021 Dec;48(4):783-811. doi: 10.1016/j.clp.2021.07.007. Epub 2021 Oct 2. PMID 34774209